CLINICAL TRIAL: NCT01442636
Title: a Prospective, Multicenter, Controlled Trial Evaluating the Implant of a Drug Eluting Stent (XIENCE PRIME, Abbott Vascular) in the Critically Ischemic Lower Leg
Brief Title: Drug Eluting Stents In The Critically Ischemic Lower Leg 2
Acronym: DESTINY 2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Flanders Medical Research Program (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMRP-101021
Record Dates: First submitted 2011-09-22; First posted 2011-09-28 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Xience Prime stent (Experimental): Patients with critical limb ischemia due to below the knee arterial lesion between 30 and 100mm in length, treated with the XIENCE PRIME™ Everolimus Eluting Coronary Stent System.
  Interventions: Device: stent

INTERVENTIONS:
Device: stent — Implantation of one or more Everolimus-eluting XIENCE PRIME™ Everolimus Eluting Coronary Stent Systems.
  Other Names: Xience Prime stent

SUMMARY:
The objective of this clinical evaluation is to evaluate the immediate and long term (up to 12 months) outcome of the XIENCE PRIME Everolimus Eluting Coronary Stent System (Abbott Vascular) in a controlled prospective investigation for the treatment of patients with critical limb ischemia due to the presence of lesions between 3cm and 10cm in length at the level of the below the knee arteries. Specifically the trial aims to illicit angiographic and ultrasound patency, clinical improvement, and adverse events associated with the use of this stent. The trial design is single armed, prospective, controlled trial run over 12 months of follow-up.

DETAILED DESCRIPTION:
The aim of this research is to evaluate the immediate and long term outcome of the XIENCE PRIME EverolimusEluting Coronary Stent System in a prospective investigation for the treatment of patients with critical limb ischemia due to the presence of lesions between 3cm and 10cm in length at the level of the below the knee arteries.

The research question is "Dose the use of an Everolimus coated stent in long tibial artery occlusions, between 3 and 10cm offer superior patency at 12 months compared to a historical cohort of bare metal stents in similar lesions?" Our hypothesis is that the use of everolimus coated stents in tibial artery occlusions between 3 and 10cm will result in lower binary restenosis than was historically found in equivalent but non-drugcoated bare metal stents.

Currently, there is evidence that angioplasty and drug eluting stents can be used as a therapy for patients with critical limb ischemia due to occlusive infrapopliteal disease. The XIENCE PRIME™ Everolimus Eluting Coronary Stent System (XIENCE PRIME EECSS or XIENCE PRIME stent system) is manufactured by Abbott. It is a device/drug combination product consisting of the CobaltChromium MULTILINK VISION 8 Coronary Stent System coated with a formulation containing everolimus, the active ingredient, embedded in a nonerodible polymer. The XIENCE PRIME Everolimus Eluting Coronary Stent is coated with everolimus (active ingredient), embedded in a nonerodible polymer (inactive ingredient). Everolimus is the active pharmaceutical ingredient in the XIENCE PRIME stent. It is a novel semisynthetic macrolide immunosuppressant, synthesized by chemical modification of rapamycin (sirolimus). The everolimus chemical name is 40O(2hydroxyethyl) rapamycin.

The XIENCE PRIME stent contains inactive ingredients including poly n-butyl methacrylate (PBMA), a polymer that adheres to the stent and drug coating, and PVDFHFP, which is comprised of vinylidene fluoride and hexafluoropropylene monomers as the drug matrix layer containing everolimus. PBMA is a homopolymer with a molecular weight (Mw) of 264,000 to 376,000 dalton. PVDFHFP is a nonerodible semicrystalline random copolymer with a molecular weight (Mw) of 254,000 to 293,000 dalton. The drug matrix copolymer is mixed with everolimus (83%/17% w/w polymer/everolimus ratio) and applied to the entire PBMA coated stent surface. The drug load is 100 μg/cm2 for all product sizes. No top-coat layer is used.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting with rest pain or minor tissue loss (Rutherford class 4 or 5)
* Patient is willing to comply with specified follow-up evaluations at the specified times
* Patient is >18 years old
* Patient understands the nature of the procedure and provides written informed consent, prior to enrolment in the study
* Patient has a projected life-expectancy of at least 12 months
* Patient is eligible for treatment with the XIENCE PRIME stent (Abbott Vascular)
* Male, infertile female, or female of child bearing potential practicing an acceptable method of birth control with a negative pregnancy test within 7 days prior to study procedure

Angiographic Inclusion Criteria:

* De novo lesion or restenotic lesion after PTA in the infrapopliteal arteries, suitable for endovascular therapy
* Total target lesion length minimally 30mm and maximally 100mm
* Target vessel diameter visually estimated to be >2.0mm and <3.5mm
* Guidewire and delivery system successfully traversed lesion

Exclusion Criteria:

* Patient refusing treatment
* The reference segment diameter is not suitable for the available stent design
* Untreated flow-limiting inflow lesions
* Perioperative unsuccessful ipsilateral percutaneous vascular procedure to treat inflow disease just prior to enrollment
* Any previous surgery in the target vessel (including prior ipsilateral crural bypass)
* Aneurysm in the target vessel
* Non-atherosclerotic disease resulting in occlusion (e.g. embolism, Buerger's disease, vasculitis)
* Severe medical comorbidities (untreated CAD/CHF, severe COPD, metastatic malignancy, dementia, etc) or other medical condition that would preclude compliance with the study protocol or 1-year life expectancy
* Major distal amputation (above the transmetatarsal) in the study limb or non-study limb
* Septicemia or bacteremia
* Any previously known coagulation disorder, including hypercoagulability
* Contraindication to anticoagulation or antiplatelet therapy
* Known allergies to stent or stent components
* Known allergy to contrast media that cannot be adequately pre-medicated prior to the study procedure
* Patient with known hypersensitivity to heparin, including those patients who have had a previous incidence of heparin-induced thrombocytopenia (HIT) type II
* Currently participating in another clinical research trial
* Angiographic evidence of intra-arterial thrombus or atheroembolism from inflow treatment
* Target lesion access not performed by transfemoral approach.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-07; Primary Completion 2013-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Primary patency at 12 months | 12 months
  Absence of restenosis (≥50% stenosis) or occlusion within the originally treated lesion based on angiography

SECONDARY OUTCOMES:
Technical success | procedure
  The ability to cross and dilate the lesion to achieve residual angiographic stenosis no greater than 30%
Hemodynamic primary patency rate at 1, 6, 12-month follow-up | 1, 6, 12-month follow-up
  Patients that present without a hemodynamically significant stenosis at the target area on duplex ultrasound (systolic velocity ratio no greater than 2.4) and without prior TLR are defined as being primary patent at the given follow-up.
Limb-salvage rate at all follow-up visits | 1, 6, 12-month follow-up
  Absence of major amputation. Major amputation is defined as amputation at or above the ankle, as opposed to minor amputation, being an amputation at or below metatarsal level, preserving functionality of the foot).
Primary assisted patency rate at 1, 6, 12-month follow-up | 1, 6, 12-month follow-up
  Defined as flow through the treated lesion maintained by repeat percutaneous intervention completed prior to complete vessel closure.
Secondary patency rate at 1, 6, 12-month follow-up | 1, 6, 12-month follow-up
  Defined as flow through the treated lesion maintained by repeat percutaneous intervention after occlusion of the target lesion.
Target lesion revascularization (TLR) at all follow-up visits | 1, 6, 12-month follow-up
  A repeat intervention to maintain or re-establish patency within the region of the treated arterial vessel plus 5 mm proximal and distal to the treated lesion edge.
Clinical success at all follow-up visits | 1, 6, 12-month
  An improvement of Rutherford classification at 1 day and 1, 6, 12-month follow-up of one class or more as compared to the pre-procedure Rutherford classification.
Serious adverse events until follow-up completions | 1,6,12 months and interim visits
  Any clinical event that is fatal, life-threatening, or judged to be severe by the investigator; resulted in persistent or significant disability; necessitated surgical or percutaneous intervention; or required prolonged hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bosiers, MD, Principal Investigator — A.Z. Sint-Blasius Hospital
Locations (6):
- Prince of Wales Private Hospital, Randwick, New South Wales, Australia
- Belgium (2):
  - Imelda Hospital, Bonheiden, Antwerp
  - Department Vascular Surgery, A.Z. Sint-Blasius Hospital, Dendermonde, East-Flanders
- Germany (3):
  - Herz-zentrum Bad Krozingen, Bad Krozingen
  - Herzzentrum, Leipzig
  - St Fransiskus hospital, Münster